CLINICAL TRIAL: NCT02805400
Title: Neurocognitive Performance During Space Flight. Validation of a Test Battery
Acronym: NeuroCog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Novespace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-A00044-45
Record Dates: First submitted 2016-04-21; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurocognitive performance (Other): Cortical activity will be determined under changing gravity level by electroencephalography (EEG/LORETA). Brain hemodynamics change will be evaluated by NIRS. Heart rate and respiratory evaluation will be indicators of cardio-vascular and central nervous arousal and stress. Cognitive performance will be evaluated by computerized tests.
  For these methods only commercially available CE marked devices will be used.
  Interventions: Other: determination of cortical activity

INTERVENTIONS:
Other: determination of cortical activity — Cortical activity will be determined under changing gravity level by electroencephalography (EEG/LORETA). Brain hemodynamics change will be evaluated by NIRS. Heart rate and respiratory evaluation will be indicators of cardio-vascular and central nervous arousal and stress. Cognitive performance will be evaluated by computerized tests.
  For these methods only commercially available CE marked devices will be used.

SUMMARY:
The main objective of this experiment is to evaluate the alterations in brain cortical activity induced by micro- and hypergravity conditions.

A secondary objective is to correlate changes in brain cortical activity and brain oxygenation level with neurocognitive performance.

Another secondary objective is to differentiate between the influences of hemodynamic and electro cortical changes and the influence of stress on cognitive performance alterations

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Persons with prior serious injuries to their head
* Persons who take any medication or drugs influencing their central nervous system or cognitive performance
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
brain cortical activity induced by micro- and hypergravity conditions : Electro cortical power in alpha frequency ranges (EEG-LORETA) | baseline
Brain tissue oxygenation ( oxy- or deoxygenated hemoglobin values) NIRS | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DP Denise, PhD, Principal Investigator — CHU CAEN
Locations (1):
- Caen CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No